CLINICAL TRIAL: NCT05487313
Title: Comparison of Pain Relief During High Thoracic Erector Spinae Plane Block Using Different Volumes of Local Anesthetics
Brief Title: Pain Relief After High Thoracic Eretor Spinae Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Hee Hong, Professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-01-026-02
Record Dates: First submitted 2022-08-01; First posted 2022-08-04 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Pain, Chronic
Keywords: Pain, Cervical, Spread
MeSH Terms: conditions — Chronic Pain; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10 ml ESP group (Active Comparator): ESP group using 10 ml mixture of local anesthetics and contrast medium
  Interventions: Procedure: Erector spinae plane block
- 20 ml ESP group (Active Comparator): ESP group using 20 ml mixture of local anesthetics and contrast medium
  Interventions: Procedure: Erector spinae plane block

INTERVENTIONS:
Procedure: Erector spinae plane block — fascial plane injection guided by fluoroscopic device after ultrasound guidance

SUMMARY:
The primary endpoint of this study was to identify if the ESPB in the patients of cervical radiculopathy has the effect of pain relief. The secondary endpoint of this study was to identify the spread level in the craniocaudal direction when performed at the T2 level.

DETAILED DESCRIPTION:
The ESPB requires ultrasound guidance which enables visible local anesthetic spread underneath the erector spinae muscles. The spinalis, longissimus thoracis, and iliocostalis muscles comprise the ES muscles, which run vertically along both sides of the vertebral column from the sacrum up to the skull base (1,10). The ESPB can be performed in the cervical, thoracic, and lumbar regions. Among them, upper or mid thoracic ESPB has been used more widely compared to cervical and lumbar regions.

Previous cadaveric studies on the ESPB at the T5 level using computed tomography (CT) reconstruction or direct dissection demonstrated the extensive craniocaudal distribution of methylene blue ranging from T1 to T8 vertebral segments deep to the ES muscles and variable involvement of epidural, paravertebral, and intercostal spaces. The ESPB performed at the T2 level of the cadaver demonstrated an injected dye distribution ranging from C4 to T10. Also, 36% of cadavers showed the spread of an injected dye to the ventral, dorsal ramus, paravertebral space, and even the contralateral side.

The exact mechanism of action of ESPB remains unclear. A recent study suggested that the analgesic effect of ESPB could be obtained by blocking the ventral and dorsal ramus of the spinal nerves by passing through the costotransverse foramen. However, in clinical practice, we can encounter highly variable clinical outcomes or sensory block after the ESPB. The study of the physical spread of the injected agent can be used to predict the clinical result and elucidate the possible mechanism of action of ESPB.

ELIGIBILITY:
Inclusion Criteria:

* cervical facet joint arthrosis
* cervical foraminal stenosis
* cervical herniated intervertebral disc
* myofascial pain syndrome of upper back muscle

Exclusion Criteria:

* Allergy to local anesthetics or contrast medium
* pregnancy
* prior history of cervical spine surgery
* coagulation abnormality

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2022-08-12 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
numerical rating scale changes among 5 times period | baseline, 10 minutes after ESPB, 1 week after ESPB, 2 weeks after ESPB, 4 weeks after ESPB, 8 weeks after ESPB
  numerical rating scale changes after T2 ESPB among 5 times period
Neck disability scale changes | baseline, 8 weeks after ESPB
  Neck disability scale changes after T2 ESPB among 2 times period

SECONDARY OUTCOMES:
spread level in the cranio-caudal direction | baseline, 1 minute after erector spinae plane block
  fluoroscopic contrast medium spread level in the cranio-caudal direction

CONTACTS AND LOCATIONS:
Overall Officials: Ji H Hong, Ph.D, Principal Investigator — Keimyung University
Locations (1):
- Hong ji HEE, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No